CLINICAL TRIAL: NCT07144488
Title: The Impact of Olive Oil Polyphenol Supplementation on Metabolic Syndrome Parameters
Brief Title: The Impact of Olive Oil Polyphenol Supplementation on Metabolic Syndrome Parameters: Preclinical Investigations Have Demonstrated That Olive Oil Polyphenols, Notably Oleocanthal, Oleacein, and Allied Secoiridoids, Possess Anti-inflammatory and Antioxidant Attributes
Acronym: OleoMetS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Apostolos Loukas Medical Centre Cyprus (Network)
Collaborators: University of Nicosia (Other); University of Crete (Other); National and Kapodistrian University of Athens (Other); Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EEBK/EP/2024/39
Record Dates: First submitted 2025-08-18; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, two-arm parallel-group study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both participants and study staff were blinded to group allocation. Placebo and active capsules were identical in appearance, weight, and taste
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olive oil aldehydic phenols (OOPs) supplement (Experimental): Participants receive a daily dose of 10 mg OOPs supplement (2 capsules, each containing 5 mg polyphenols). The formulation consists of 75% oleocanthal/oleacein and 25% oleuropein aglycon/ligstroside aglycon.
  Interventions: Dietary Supplement: Olive Oil Polyphenol Supplement (OOPs, OLEOPROTECT®, Thousand Olives®)
- Placebo supplement (Placebo Comparator): Participants receive 2 placebo capsules daily, identical in weight, appearance, and taste to the active supplement. Placebo contains PEG400, cellulose, silicon dioxide, and magnesium stearate, but no active olive oil polyphenols.
  Interventions: Dietary Supplement: Placebo capsules

INTERVENTIONS:
Dietary Supplement: Olive Oil Polyphenol Supplement (OOPs, OLEOPROTECT®, Thousand Olives®) — Participants receive two capsules daily (total 10 mg/day) of a standardized olive oil polyphenol extract. Each capsule contains 5 mg of aldehydic phenols: 75% oleocanthal/oleacein and 25% oleuropein aglycon/ligstroside aglycon. Formulated with PEG400, cellulose, silicon dioxide, and magnesium stearate. Duration: 12 weeks.
  Other Names: Olive oil aldehydic phenols (OOPs) supplement
  Arms: Olive oil aldehydic phenols (OOPs) supplement
Dietary Supplement: Placebo capsules — Two capsules taken daily for 12 weeks. Identical in weight, appearance, and taste to the active OOPs capsules. Contain PEG400, cellulose, silicon dioxide, and magnesium stearate, but no active olive oil polyphenols.
  Arms: Placebo supplement

SUMMARY:
Olive oil polyphenols, particularly oleocanthal, oleacein, and related secoiridoids, have shown anti-inflammatory and antioxidant properties in preclinical studies. Metabolic syndrome (MetS) is characterized by a constellation of risk factors, including central obesity, dyslipidemia, hypertension, and dysglycemia, which collectively contribute to a substantially elevated risk of cardiovascular disease (CVD) and type 2 diabetes mellitus (T2DM). Preclinical investigations have demonstrated that olive oil polyphenols, notably oleocanthal, oleacein, and allied secoiridoids, possess anti-inflammatory and antioxidant attributes.

The goal of this clinical trial is to learn if a polyphenol-rich olive oil extract works to improve metabolic syndrome (MetS) parameters in adults. It will also evaluate the safety of the supplement. The main questions it aims to answer are:

Does the olive oil extract improve fasting blood glucose and HbA1c levels?

How does the supplement affect other health measures such as cholesterol levels, inflammation (CRP), body mass index (BMI), blood pressure, waist size, liver function (ALT), kidney function (eGFR), uric acid levels, and fatigue?

Researchers will compare the olive oil extract supplement to a placebo (a look-alike substance with no active ingredients) to see if the supplement can help manage metabolic syndrome.

Participants will:

Take either 10 mg of the olive oil extract supplement or a placebo once daily for 12 weeks

Attend clinic visits for tests and checkups at the beginning and end of the study period

Have their blood sugar, cholesterol, inflammation markers, liver and kidney function, and other health parameters measured before and after the treatment

Complete questionnaires assessing fatigue levels

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 30-70 years with a diagnosis of MetS per International Diabetes Federation criteria were enrolled after informed consent.

Exclusion Criteria:

-

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Glycated haemoglobin | 12 weeks
  Change in HbA1c levels
Fasting blood glucose | 12 weeks
  Change in fasting blood glucose levels

SECONDARY OUTCOMES:
Lipid profile | 12 weeks
  Change in HDL, LDL, total cholesterol, triglycerides (mg/dL) and oxidised LDL
Fatigue / Energy levels | 12 weeks
  Change from baseline in fatigue scores measured by the Energy Level Questionnaire (ELQ), which includes general, physical, and mental fatigue subscales. Each item is scored on a 5-point scale: Not at all, A little, Moderately, Quite a bit, Very much. Higher scores indicate greater fatigue (worse outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Apostolos Loukas Medical Centre Cyprus, Nicosia, Engomi, Cyprus

REFERENCES:
- [Derived] Samoutis G, Kyriakides TC, Demetriou N, Poulianiti E, Samouti G, Samouti S, Diamantakos P, Melliou E, Magiatis P. The impact of olive oil polyphenol supplementation on metabolic syndrome parameters The OleoMetS study: A randomized, controlled clinical trial. Clin Nutr ESPEN. 2025 Dec 20;71:102883. doi: 10.1016/j.clnesp.2025.102883. Online ahead of print. PMID 41429309